CLINICAL TRIAL: NCT00841490
Title: Oral H. Pylori Prevalence in Intellectually & Developmentally Disabled Adults
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Catherine J Binkley, Associate Professor, University of Louisville
Other Study IDs: OGMB080062; 1R21DE017378-01A2 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2016-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Oral Health; Intellectually & Developmentally Disabled

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of dental plaque.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Intellectually & Developmentally Disabled Adults
- 2: Control Group of Adults without Intellectual & Developmental Disabilities

SUMMARY:
The purpose of this study is to determine if the bacteria that cause gastric infections can be found in the mouths of intellectually and developmentally disabled persons. If the bacteria that causes gastric infections is found in the mouth it may be swallowed and contribute to gastric infections.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) bacteria play a significant role in the etiology of gastric and duodenal ulcers, gastro-esophageal reflux disease and gastric adenocarcinoma. Intellectually disabled/developmentally disabled (ID/DD) adults are reported to have H. pylori infection at approximately twice the rate of the general population and experience recurrence at a seven-fold higher rate, contributing to increased mortality due to gastric cancer. The oral cavity may serve as a reservoir for H. pylori and subsequently contribute to the recurrence of gastric infection.

Numerous studies have identified H. pylori in dental plaque, an environment that is relatively resistant to systemic antibiotics. Systemic antibiotics are used to treat H. pylori infections but do not appear to eradicate H. pylori in the mouth. The oral status of ID/DD adults is reported to be poor due to inadequate oral hygiene, leading to increased plaque, caries and periodontal disease. Furthermore, poor oral status (periodontal disease) has been associated with H. pylori seropositivity. While ID/DD adults have elevated rates of H. pylori gastric infections, nothing is known about the prevalence of H. pylori in their oral cavities.

The proposed exploratory research will address the following questions in this disadvantaged population: 1) What is the prevalence of H. pylori in the dental plaque in ID/DD adults?, 2) Is poor oral status associated with H. pylori gastric infection?, and 3) Does H. pylori persist in the dental plaque of ID/DD adults after systemic antibiotic treatment, and if so, is it associated with recurrence of gastric infection? This epidemiological study of 112 institutionalized ID/DD and 112 control subjects will involve oral examinations, indices, dental plaque sampling, and C13 Urea Breath Tests at baseline to determine prevalence. Nested Polymerase Chain Reaction (PCR) analyses will be used to detect H. pylori in the dental plaque. For those ID/DD subjects who have a positive gastric H. pylori test at baseline, repeated oral sampling and gastric tests will be performed over 1 year to determine persistence.

If poor oral health status and oral H. pylori prevalence are correlated with gastric H. pylori infections, a future pilot clinical trial will be conducted to investigate the concordance between genetic strains of H. pylori in the mouth and stomach, the effect of various interventions on oral health, oral H. pylori prevalence, and H. pylori gastric infections in ID/DD adults. The proposed research responds to the Surgeon General's National Call to Action to conduct studies to elucidate underlying mechanisms and determine any causal associations between oral infections and systemic conditions. The proposed research also addresses the need to reduce health disparities, improve quality of life, and reduce morbidity and mortality in vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

ID/DD participants:

1. Mild, moderate, or severe intellectual and/or developmental disability (IQ < 50).
2. Dependent in two or more Activities of Daily Living.\
3. Unable to perform adequate oral hygiene.
4. At least six teeth present in the oral cavity including 6 posterior teeth present

Control Group Participants:

1. At least 6 posterior teeth present, and
2. Age and gender match to an ID/DD subject.

Exclusion Criteria (Both Groups):

1. Antibiotics taken 2 weeks prior to baseline.
2. Proton pump inhibitors taken 2 weeks prior to baseline.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A study involving 110 intellectually disabled and/or developmentally disabled (ID/DD) participants aged 18 to 90 years of age at a facility in Kentucky will be conducted. An age and gender matched control group (n = 110) will also be evaluated for oral H. pylori prevalence and H. pylori gastric infections. The control group will be recruited and enrolled from the general dental clinics at the University of Louisville School of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of H. pylori in dental plaque | one year

SECONDARY OUTCOMES:
Association of oral health status and/or oral H. pylori with H. pylori gastric infection | one year
Persistence of H. pylori in the dental plaque of ID/DD adults after systemic antibiotic treatment | one year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Binkley, DDS, PhD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - University of Louisville School of Dentistry, Louisville, Kentucky
  - Bluegrass Oakwood, Somerset, Kentucky

IPD SHARING:
Plan to Share IPD: No